CLINICAL TRIAL: NCT06064890
Title: A Phase 1/2 Open-Label, Ascending Dose, Multicenter Study to Evaluate the Safety and Preliminary Efficacy of AVB-101 Administered by Bilateral Intrathalamic Infusion in Subjects With Frontotemporal Dementia With Progranulin Mutations (FTD-GRN)
Brief Title: A Study to Evaluate the Safety and Effect of AVB-101, a Gene Therapy Product, in Subjects With a Genetic Sub-type of Frontotemporal Dementia (FTD-GRN)
Acronym: ASPIRE-FTD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AviadoBio Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AVB-PGRN-001; 2023-509444-10-00 (EU CTIS Number)
Record Dates: First submitted 2023-09-12; First posted 2023-10-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Frontotemporal Dementia; FTD; FTD-GRN; Dementia, Frontotemporal
Keywords: Gene Therapy; AAV; Intrathalamic; Intraparenchymal; Progranulin; Behavioral Variant FTD; Primary Progressive Aphasia; PGRN; Granulin; Dementia; Dementia Gene Therapy; AAV9
MeSH Terms: conditions — Frontotemporal Dementia; Aphasia, Primary Progressive; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Cohort 1 (dose 1) (Experimental): Initial dose, delivered as a one-time only, intrathalamic administration.
  Interventions: Procedure: Intrathalamic AAV.PGRN administration; Genetic: Intrathalamic AVB-101
- Cohort 2 (dose 2) (Experimental): Escalated dose, delivered as a one-time only, intrathalamic administration.
  Interventions: Procedure: Intrathalamic AAV.PGRN administration; Genetic: Intrathalamic AVB-101
- Cohort 3 (dose 3) (Experimental): Additional dose, delivered as a one-time only, Intrathalamic administration.
  Interventions: Procedure: Intrathalamic AAV.PGRN administration; Genetic: Intrathalamic AVB-101

INTERVENTIONS:
Procedure: Intrathalamic AAV.PGRN administration — One-time MRI-guided stereotaxic infusion of AAV.PGRN into the brain
Genetic: Intrathalamic AVB-101 — AVB-101 is made from an adeno-associated virus, serotype 9 (AAV9). AAVs are small viruses that are naturally occurring and do not cause illness or infection on their own. AVB-101 has been modified to contain a copy of the correct (non-mutated) GRN gene, plus some other genetic material to enable the GRN gene to function inside neurons (cells within the brain). AVB-101 has also been modified so that it cannot divide and make new copies of itself (known as 'replication'), which means that it cannot cause disease or a large immune response in your body.

SUMMARY:
The goal of this clinical study is to learn about an investigational gene therapy product called AVB-101, which is designed to treat a disease called Frontotemporal Dementia with Progranulin Mutations (FTD-GRN). FTD-GRN is an early-onset form of dementia, a progressive brain disorder that affects behavior, language and movement. These symptoms result from below normal levels of a protein called progranulin (PGRN) in the brain, which leads to the death of nerve cells (neurons), affecting the brain's ability to function.

The main questions that the study aims to answer are:

1. Is a one-time treatment with AVB-101 safe for patients with FTD-GRN?
2. Does a one-time treatment with AVB-101 restore PGRN levels to at least normal levels?
3. Could AVB-101 work as a treatment to slow down or stop progression of FTD-GRN?

In this study there is no placebo (a dummy pill or treatment used for comparison purposes), so all participants will receive a one-time treatment of AVB-101 delivered directly to the brain, with follow-up assessments for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 30 to 75 years of age
* Carriers of a pathogenic GRN mutation
* FTD as evidenced by CDR + NACC FTLD global score of 0.5, 1.0, or 2.0
* Presence of 1 or more of the criteria for diagnosis of possible bvFTD or PPA
* Able and willing to comply with all procedures and the study visit schedule
* Able and willing to give written informed consent prior to study participation, and agree to designate a legal representative to act on their wishes to continue participation should they lose capacity to consent at some point during the study OR If, in the Investigator's opinion, the subject lacks capacity to consent, written informed consent of their legal representative must be obtained in accordance with local laws, regulations, and/or customs. In countries where local laws, regulations, and/or customs do not permit subjects who lack capacity to consent to participate in this study, these subjects will not be enrolled
* An identified, informed study partner who is able and willing to support the participant in the study and to provide assessments of the participant during the study

Exclusion Criteria:

* Severe dementia, defined as CDR + NACC FTLD global score of 3.0, or other symptoms that preclude the ability to comply with study procedures and/or pose unacceptable safety risk to the subject
* Any concurrent disease that may cause cognitive impairment unrelated to mutations in the GRN gene, such as other causes of dementia, neurosyphilis, hydrocephalus, stroke, small vessel ischemic disease, uncontrolled hypothyroidism, or vitamin B12 deficiency
* Clinically significant abnormality on MRI at Screening considered to be a contraindication to Intrathalamic infusion
* Surgically significant pattern of brain atrophy on MRI at Screening that interferes with planned neurosurgical trajectory
* Previous treatment with any gene or cell therapy
* Previous treatment with any investigational medicinal product (IMP) within 60 days or 5 half-lives (whichever is longer) prior to study drug treatment
* Concomitant disease, any clinically significant laboratory abnormality, or treatment which, in the opinion of the Investigator, may pose an unacceptable safety risk to the participant or interfere with study conduct or the participant's ability to comply with study procedures including neurosurgical administration under anesthesia

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2030-03-21 (Estimated)

PRIMARY OUTCOMES:
Number and incidence of AEs and SAEs | Up to week 26
  Type and incidence of adverse events
Change from baseline in the Mini-Mental State Examination (MMSE) | Up to week 12
  Mini-Mental State Examination (MMSE) is a global assessment of cognitive status. Score range 0-30; higher scores reflect better cognitive function. Change in MMSE score from baseline visit to post-treatment visit will be assessed.
Incidence of treatment emergent suicidal ideation or behavior | 26 week initial, 5-year total follow-up period
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is an assessment tool that evaluates suicidal ideation and behavior. C-SSRS will be measured at each visit to assess for absence/presence of suicidal ideation and/or behavior.
Incidence of treatment-emergent clinically significant abnormalities in clinical examination findings | 5-year total follow-up period
Incidence of treatment-emergent clinically significant abnormalities in safety laboratory values | 5-year total follow-up period
Change from baseline in brain structure | 5-year total follow-up period
  Assessed by presence of any clinically significant MRI findings at post treatment visits including brain swelling or bleeding

SECONDARY OUTCOMES:
Change from baseline in PGRN protein levels in CSF and blood | 26-week initial and 5-year total follow-up period
  Change over time in level of PGRN
Change from baseline in NfL levels in CSF and blood | 26-week initial and 5-year total follow-up period
  Change over time in level of NfL
Change from baseline in CDR + NACC FTLD-SB score | 5-year total follow-up period
  The Clinical Dementia Staging Instrument (CDR) plus National Alzheimer's Coordinating Center Frontotemporal Degeneration domains (NACC FTLD) was developed as a way to improve characterization of cognitive and global function in patients with FTLD. The CDR+NACC FTLD score will capture patients' disease status. CDR+NACC FTLD Sum of Boxes (SB) score refers to the sum of the scores of each domain (sum of boxes) that ranges from 0 to 24.
Time to achieve clearance of vector genomes | Up to week 26
  Measured in plasma and semen (males only)
Change from baseline in brain volumes | 5-year total follow-up period
  Calculation based upon 3DT1 MRI scans
Change from baseline in AAV9 immunogenicity in blood | 5-year total follow-up period
  Measured by level of antibodies and ELISPOT to AAV9 capsid
Change from baseline in AAV9 immunogenicity in CSF | 5-year total follow-up period
  Measured by level of antibodies to AAV9 capsid
Change from baseline in PGRN immunogenicity in CSF | 5-year total follow-up period
  Measured by level of antibodies to PGRN protein
Change from baseline in PGRN immunogenicity in blood | 5-year total follow-up period
  Measured by level of antibodies and ELISPOT to PGRN protein
Change in Caregiver Global Impression of Change (CaGI-C) | 5-year total follow-up period
  Global impression of change as assessed by the caregiver. The CaGI-C is a 7 point scale where 1= very much improved, 7= very much worse.
Change in Patient Global Impression of Change (PGI-C) | 5-year total follow-up period
  Global impression of change as assessed by the patient. The PGI-C is a 7 point scale where 1= very much improved, 7= very much worse.
Change in Clinical Global Impression of Change (CGI-C) | 5-year total follow-up period
  Global impression of change as assessed by the investigator (clinician). The CGI-C is a 7 point scale where 1= very much improved, 7= very much worse.
Change from baseline in GRN-specific Genetic Frontotemporal Initiative Cognitive (GENFI-Cog) composite score | 5-year total follow-up period
  Calculated from the neuropsychological test battery that assesses various cognitive domains: language, attention/processing speed, executive function, verbal and visuospatial memory and social cognition.
  Scores from the neuropsychological test battery are converted using standard statistical methods into the composite score. The GRN specific composite score is expected to be more sensitive to detect changes in cognition that are associated with FTD, and will be compared to the baseline score. Lower scores indicate worse performance.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (3):
  - The Ohio State University (OSU) Wexner Medical Center, Columbus, Ohio
  - Vanderbilt University Medical Centre, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy
- Amsterdam UMC, Amsterdam, Netherlands
- Poland (6):
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Katowice
  - Neurologia Slaska Centrum Medyczne, Katowice
  - Uniwersyteckie Centrum Kliniczne, SUM w Katowicach, Katowice
  - Euromedis Sp. z o.o., Szczecin
  - Centrum Medyczne NeuroProtect Sp z o.o., Warsaw
  - Mazowiecki Szpital Brodnowski Sp. z o. o., Warsaw
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitari i Politecnic La Fe, Valencia
- Skåne University Hospital, Lund, Sweden
- United Kingdom (3):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - University Hospital of Wales, Cardiff
  - University College London Hospitals, London

IPD SHARING:
Plan to Share IPD: No